CLINICAL TRIAL: NCT05973981
Title: The Impact of Standardized Tobacco Product Packaging on Young Adults in the Retail Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01CA261639 (NIH)
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Status Quo Packages (Active Comparator): Cigarette packages appear as they normally do - no standardization
  Interventions: Behavioral: Package standardization
- Partial standardization (Experimental): Cigarette packages appear with half of the package using a standardized color
  Interventions: Behavioral: Package standardization
- Full standardization (Experimental): Cigarette packages appear with all of the packages fully standardized (by color and font)
  Interventions: Behavioral: Package standardization

INTERVENTIONS:
Behavioral: Package standardization — Conditions vary in terms of amount of cigarette packages that are subject to standardization

SUMMARY:
The overall aim of this research is to experimentally evaluate the extent to which partially standardizing the color of tobacco packaging influences tobacco use intentions among young adults who have varying levels of tobacco use experience.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-34
* Past month cigarette smoker

Exclusion Criteria:

* None.

Ages: 21 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 433 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RAND Corporation, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Status Quo Packages | Partial Standardization | Full Standardization
Started | 143 | 143 | 147
Completed | 143 | 143 | 147
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Status Quo Packages | Partial Standardization | Full Standardization | Total
Number analyzed (Participants) | 143 | 143 | 147 | 433
Age, Customized [Count of Participants; unit: Participants]
  Age group: 21-25 | 85 | 79 | 79 | 243
  Age group: 26-34 | 57 | 63 | 68 | 188
  Age group: missing | 1 | 1 | 0 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 68 | 62 | 68 | 198
  Male | 59 | 67 | 62 | 188
  other endorsed | 16 | 14 | 17 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 9 | 24
  Not Hispanic or Latino | 134 | 136 | 138 | 408
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 52 | 48 | 46 | 146
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 19 | 25 | 59
  White | 54 | 62 | 55 | 171
  More than one race | 13 | 9 | 11 | 33
  Unknown or Not Reported | 9 | 5 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Quit Smoking Motivation
Description: Motivation to quit smoking as assessed by the Motivation to Stop Scale (MTSS; Kotz et al., 2013; Drug and Alcohol Dependence) participants endorsing one of 7 items:
  1. = I don't want to stop smoking.
  2. = I think I should stop smoking but don't really want to.
  3. = I want to stop smoking but haven't thought about when.
  4. = I REALLY want to stop smoking but I don't know when I will.
  5. = I want to stop smoking and hope to soon.
  6. = I REALLY want to stop smoking and intend to in the next 3 months.
  7. = I REALLY want to stop smoking and intend to in the next month.
Time Frame: Immediately after shopping in the RAND StoreLab
Population: Two participants are missing data on the outcome - they declined to respond to the item.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Status Quo Packages | Partial Standardization | Full Standardization
Number analyzed (Participants) | 143 | 141 | 147
score on a scale | 3.7 [3.4 to 4.0] | 3.9 [3.6 to 4.2] | 3.7 [3.4 to 4.0]
Statistical Analysis 1: Comparison: Status Quo Packages vs Partial Standardization; Test type: Other; Slope = 0.19, 95% CI 2-sided [-0.25 to 0.63] — Adjusted for age, sex, and race
Statistical Analysis 2: Comparison: Status Quo Packages vs Full Standardization; Test type: Other; Slope = 0.03, 95% CI 2-sided [-0.41 to 0.46] — adjusted for age, sex, and race

ADVERSE EVENTS:
Time Frame: Immediate, day of session
Arm/Group | Status Quo Packages | Partial Standardization | Full Standardization
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/143 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/143 | 0/147
Other Adverse Events (participants affected / at risk) | 0/143 | 0/143 | 0/147

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT05973981/Prot_SAP_000.pdf